CLINICAL TRIAL: NCT07326800
Title: Efficacy of the MAEva Program (Meditation, Acceptance, and Commitment to Values) in Breast Cancer Patients Undergoing Chemotherapy : a Randomized, Multicenter Clinical Trial
Brief Title: Efficacy of the MAEva Program (Meditation, Acceptance, and Commitment to Values) in Breast Cancer Patients Undergoing Chemotherapy
Acronym: MAEva-MCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-A01424-45
Record Dates: First submitted 2025-09-09; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Non Metastatic Breast Cancer; Chemotherapy
Keywords: Cancer; MAEva program; Mindfulness; Acceptance and commitment therapy; Quality of life
MeSH Terms: conditions — Neoplasms | interventions — Meditation; Perceived Stress Scale; Patient Health Questionnaire

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAEva program group (Experimental): The MAEva program is an open group intervention (i.e., patients can enter the program at any session), and it is circular (i.e., it is possible to do the three sessions in any order and repeat the program to benefit from a training effect). Patients are invited to participate according to their possibilities and without having to commit to carrying out the whole program (i.e., it is fully acceptable for a patient to participate in only one or two of the three sessions of a complete cycle).
  Patients will be able to participate in one weekly session for nine consecutive weeks.
  Interventions: Other: MAEva program (Meditation, Acceptance and Commitment to Values or "Méditation, Acceptation et Engagements en direction des valeurs")
- Discussion group (Active Comparator): The discussion group is structured according to the same schedule as MAEva program. It is an open group intervention (i.e., patients can enter at any session), and it is circular (i.e., it is possible to do the three sessions in any order and repeat the program to benefit from a training effect). Patients are invited to participate according to their possibilities and without having to commit to carrying out the whole program (i.e., it is fully acceptable for a patient to participate in only one or two of the three sessions of a complete cycle).
  Patients will be able to participate in one weekly session for nine consecutive weeks.
  Interventions: Other: Discussion group

INTERVENTIONS:
Other: MAEva program (Meditation, Acceptance and Commitment to Values or "Méditation, Acceptation et Engagements en direction des valeurs") — MAEva program combines ACT and mindfulness practices, and comprises three group sessions of 1 h 30 min each, following a weekly schedule. Each session addresses a specific theme and contains short meditative practices (10-15 min), as well as sharing times with feedback of experience and theoretical contributions: Session 1: Mindfulness Meditation (targeted processes: contact with the present moment and self-as-context), Session 2: Acceptance (targeted processes: acceptance and defusion), and Session 3: Commitment to Values (targeted processes: values and committed action).
  Between sessions, participants were encouraged to engage in daily practice of the ACT therapeutic processes covered. Moreover, they were invited to cultivate mindfulness in daily life through informal exercises, that is, to devote oneself attentively to routine activities.
  Other Names: Perceived Stress Scale; Anxiety and/or depression; Quality of life evaluations (Quality of Life Questionnaire, Breast Cancer module, Fatigue); Multidimensional Psychological Flexibility Inventory; Satisfaction questionnaire and semi-structured interview
  Arms: MAEva program group
Other: Discussion group — Discussion group comprises three group sessions of 1 h 30 min each, following a weekly schedule. Each session addresses a specific theme : Session 1: Treatments, Session 2: Fatigue, and Session 3: Social life.
  The facilitators will limit themselves to supportive interview techniques (listening, open-ended questions, rephrasing, expressing empathy) and, if necessary, will refer participants to the resources available at each center.
  Other Names: Perceived Stress Scale; Anxiety and/or depression; Quality of life evaluations (Quality of Life Questionnaire, Breast Cancer module, Fatigue); Multidimensional Psychological Flexibility Inventory; Satisfaction questionnaire and semi-structured interview
  Arms: Discussion group

SUMMARY:
The MAEva program combines Acceptance and Committment Therapy (ACT) and mindfulness practices. It is an open and circular intervention, in three sessions (Mindfulness, Acceptance, and Commitment to values). It is designed for cancer patients and was the subject of an initial study that explored its feasibility and acceptability, as well as the initial results on psychological well-being.

This randomized, multicenter clinical trial is necessary to demonstrate the efficacy of the MAEva program compared to a discussion group with non metastatic breast cancer patients undergoing chemotherapy.

Patients will be included and randomized into two arms:

* In the first arm, patients will have the opportunity to participate in the MAEva program for nine consecutive weeks.
* and the second arm patients will have the opportunity to participate in a discussion group for nine consecutive weeks.

The patients will be able to attend one session per week for nine consecutive weeks.

Quantitative assessments of quality of life, symptoms of stress, anxiety, and depression, as well as psychological flexibility, will be conducted before the first session, after 3 weeks, 9 weeks, and 12 weeks.

Also, a qualitative analysis will be conducted based on satisfaction questionnaire and a semistructured interview performed after the end of the program. The interview analysis will described the extent to which the intervention is adapted to the realities on the ground and the needs of the target population. It will enable to identify how patients appropriate the psychological flexibility processes taught in the program in relation to the conceptual framework of ACT therapy (i.e., contact with the present moment, self-as-context, acceptance, defusion, values, and committed action) and integrate them into their daily lives.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-metastatic breast cancer currently undergoing chemotherapy,
* Patients who are able and willing to follow all study procedures in accordance with the protocol,
* Patients who have understood, signed, and dated the consent form,
* Patients who are affiliated with the social security system,
* Patients who are able to remain seated during the 1.5-hour sessions.

Exclusion Criteria:

* Patients with metastatic cancer,
* Presence of an acute psychiatric disorder: acute depression, unstable bipolar disorder, psychotic disorder (delusions, hallucinations), etc.
* Presence of recurrent uncontrolled panic attacks (particularly related to hypochondriacal concerns),
* Insufficient attentional resources for meditation: major attention, memory, or reasoning disorders,
* Presence of cognitive and neurocognitive disorders and deficits,
* Presence of deafness,
* Current participation in another mindfulness program,
* Persons deprived of their liberty or under guardianship (including curatorship),
* Inability to undergo medical monitoring for the trial for geographical, social, or psychological reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 190 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the efficacy of the MAEva program versus discussion group on quality of life in patients with non-metastatic breast cancer undergoing chemotherapy. | At 12 weeks after first session
  Evolution in the overall QLQ-C30 quality of life (QoL) score at 12 weeks compared to a control group.
  Different dimensions of quality of life will be assessed using the EORTC QLQ-C30 (QoL Questionnaire); It includes five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high / healthy level of functioning, A high score for the global health status / QoL represents a high QoL, A high score for a symptom scale / item represents a high level of symptomatology / problems.

SECONDARY OUTCOMES:
the MAEva program's efficacy on stress symptoms | From enrollement at 12 weeks after first session
  Improvement in symptoms of stress compared to a control group. Stress will be assessed using the Perceived Stress Scale (PSS-10).
the MAEva program's efficacy on symptoms of anxiety and depression (identification of a cut-off level for anxiety and depression) | From enrollment at 12 weeks after first session
  Improvement in symptoms of anxiety, and depression compared to a control group. Anxiety and/or depression will be assessed using the Hospital Anxiety and Depression Scale (HADS).
the MAEva program's efficacy on different dimensions of quality of life | From enrollment at 12 weeks after first session
  Assessement of quality of life compared to a control group. Different dimensions of quality of life will be assessed using the EORTC QLQ-C30 (Quality of Life Questionnaire); It includes five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status / QoL scale.
the MAEva program's efficacy on quality of life in breast cancer patients | From enrollment at 12 weeks after first session
  Assessement of quality of life compared to a control group. Quality of life in breast cancer patients will be assessed using the EORTC-BR23 (Breast Cancer module); it includes five multi-item scales to assess body image, sexual functioning, systemic therapy side effects, breast symptoms, and arm symptoms.
the MAEva program's efficacy on fatigue | From enrollment at 12 weeks after first session
  Assessement of quality of life compared to a control group. Fatigue will be assessed using the EORTC-FA12 (Fatigue); It includes three multi-item scales to assess physical fatigue, emotional fatigue, and cognitive fatigue.
the MAEva program's efficacy on Psychological Flexibility | From enrollment at 12 weeks after first session
  Assessment of psychological flexibility (Multidimensional Inventory of Psychological Flexibility (MPFI-24))
the MAEva program's efficacy on the psychological processes involved in acceptance and commitment therapy | At 12 weeks after first session
  Assessment of processes (i.e., contact with the present moment, self-as-context, acceptance, defusion, values, and committed action) at play during the intervention (semi-structured interviews (qualitative analysis))
Adherence | From enrollment at 9 weeks after first session
  Patient participation rate.
Assessement of Satisfaction | At 12 weeks after first session
  Assessment of patient satisfaction (subjective score between 1 and 10; open-ended questions (qualitative analysis)) Assessment of caregiver satisfaction (subjective score between 1 and 10; open-ended questions (qualitative analysis))

CONTACTS AND LOCATIONS:
Overall Officials: François Bourgognon, MD, Principal Investigator — Institut de Cancérologie de Lorraine; Denise BECHET, PhD, Study Chair — Institut de Cancérologie de Lorraine

REFERENCES:
- [Background] Bourgognon F, Bechet D, Huin-Schohn C, Strelow A, Demarche L, Guillou M, Adam V, Fall E, Omorou AY. A mixed method feasibility and acceptability study of a flexible intervention based on acceptance and commitment therapy for patients with cancer. Front Psychol. 2024 Jul 3;15:1409308. doi: 10.3389/fpsyg.2024.1409308. eCollection 2024. PMID 39021646